CLINICAL TRIAL: NCT00502242
Title: A Randomized, Placebo Controlled, Double-Blind Comparative Study Evaluating The Effect of Ramipril On Urinary Protein Excretion In Maintenance Renal Transplant Patients Converted To Sirolimus
Brief Title: Study Evaluating The Effect Of Ramipril On Urinary Protein Excretion In Renal Transplant Patients Converted To Sirolimus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0468E5-4439; B1741001
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Capsule - initial treatment is 5 mg (active)- oral - once per day
  Interventions: Drug: ramipril
- B (Placebo Comparator): Capsule - initial treatment is 5 mg (placebo) - oral - once per day
  Interventions: Drug: ramipril

INTERVENTIONS:
Drug: ramipril — Capsule - initial treatment is 5 mg (active)- oral - once per day
  Arms: A
Drug: ramipril — Capsule - initial treatment is 5 mg (placebo) - oral - once per day
  Arms: B

SUMMARY:
The primary objective of the study is to determine the efficacy of ramipril in preventing a urinary protein to creatinine ratio (U p/c) greater than 0.5 following conversion to sirolimus from a calcineurin inhibitor (CNI) in maintenance kidney transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Receiving cyclosporine (CsA) or tacrolimus (TAC) since the first month post-transplant.
* In addition to a calcineurin inhibitor (CNI), subjects must be treated with either corticosteroids at a dosage range of 2.5 to 15 mg/day for prednisone or prednisolone (2 to 12mg/day for methylprednisolone or the alternate day equivalent) or a steroid-free regimen for a minimum of 12 weeks before randomization or either MMF (>/=500mg/day), mycophenolate sodium (MPS) (>/=360 mg/day) or AZA (>/=50mg/day). Subjects must be taking a minimum of 2 immunosuppressive drugs if on a steroid-free regimen.
* Subject is 3 to 60 months after renal transplantation.
* Subject is greater than 12 weeks after treatment for any acute rejection.

Exclusion Criteria:

* Subjects who are currently receiving, or have received within 4 weeks before enrollment, RAAS blockade.
* Subjects with a calculated GFR < 40mL/min (per the Modification of Diet in Renal Disease [MDRD-7] or abbreviated MDRD formula).
* Subjects with a urine protein to creatinine ratio (U p/c) of >0.3.
* Subjects with a history of uncontrolled systolic blood pressure (SBP >140 mm Hg).
* Subjects with severe hepatic impairment (Grade C Child-Pugh score). Additional Inclusion / Exclusion Criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2007-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- United States (19):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Portland, Maine
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, Gosse Pointe, Michigan
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Valhalla, New York
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Harrisburg, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
- Argentina (4):
  - Pfizer Investigational Site, Capital Federal, Buenos Aires
  - Pfizer Investigational Site, San Martín, Buenos Aires
  - Pfizer Investigational Site, Buenos Aires
  - Pfizer Investigational Site, Córdoba
- Australia (3):
  - Pfizer Investigational Site, Brisbane, Queensland
  - Pfizer Investigational Site, North Terrace
  - Pfizer Investigational Site, Woodville South
- Pfizer Investigational Site, Linz, Austria
- Brazil (3):
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Pfizer Investigational Site, Montreal, Quebec, Canada
- Pfizer Investigational Site, Erlangen, Germany
- Pfizer Investigational Site, Szeged, Hungary
- Pfizer Investigational Site, Petah Tikva, Israel
- Mexico (2):
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Veracruz, Mexico
- Pfizer Investigational Site, Szczecin, Poland
- South Africa (2):
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Cape Town, Western Cape

REFERENCES:
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471
- [Derived] Mandelbrot DA, Alberu J, Barama A, Marder BA, Silva HT Jr, Flechner SM, Flynn A, Healy C, Li H, Tortorici MA, Schulman SL. Effect of Ramipril on Urinary Protein Excretion in Maintenance Renal Transplant Patients Converted to Sirolimus. Am J Transplant. 2015 Dec;15(12):3174-84. doi: 10.1111/ajt.13384. Epub 2015 Jul 14. PMID 26176342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Randomized, Placebo Controlled, Double-Blind Comparative Study Evaluating the Effect of Ramipril on Urinary Protein Excretion in Maintenance Renal Transplant Patients Converted to Sirolimus.
Pre-assignment Details: Eligible participants were randomly assigned in a Double-Blind fashion to the Ramipril treatment group or the Placebo control group.
Groups:
- Ramipril: Participants were receiving cyclosporine (CsA) or tacrolimus (TAC) and either mycophenolate mofetil (MMF), mycophenolate sodium (MPS), or azathioprine (AZA) or steroids dosed per center's standard of care. Participants received ramipril, 5 or 10 milligrams per day (mg/d) orally (PO). 2-6 weeks after randomization, participants stopped TAC or CsA (within 21 days of sirolimus [SRL] initiation) and received SRL, PO, 2-4 mg/d (6-12 mg on Day 1 if TAC or CsA withdrawn abruptly) to achieve target trough levels (7-15 nanograms per milliliter [ng/mL] less than [<]1 year post-transplant [PT], 5-15 ng/mL greater than or equal to [≥]1 year PT) for up to 52 weeks. Ramipril was increased to 10-20 mg if urinary protein to creatinine ratio (U p/c) was ≥0.5. If U p/c ≥0.5 persisted, losartan 50 mg/d was added; if U p/c ≥0.5 still persisted, losartan was increased to 100 mg/d. If then U p/c <0.5 was not maintained, study medication was discontinued and participant entered off-therapy phase of study.
- Placebo: Participants were receiving CsA or TAC and either MMF, MPS, or AZA or steroids dosed per center's standard of care. Participants received double-blinded placebo, 1 capsule (5 or 10 mg/day), PO. 2-6 weeks after randomization, participants stopped TAC or CsA (within 21 days of SRL initiation) and received SRL, PO, 2-4 mg/d (6-12 mg on Day 1 if TAC or CsA withdrawn abruptly) to achieve target trough levels (7-15 ng/mL <1 year PT, 5-15 ng/mL ≥1 year PT) for up to 52 weeks. Placebo dose was doubled if U p/c was ≥0.5. If U p/c ≥0.5 persisted, losartan 50 mg/d was added; if U p/c ≥0.5 still persisted, losartan was increased to 100 mg/d. If then U p/c <0.5 was not maintained, study medication was discontinued and participant entered off-therapy phase of study.
Period: Overall Study
Arm/Group | Ramipril | Placebo
Started | 155 | 140
Completed | 104 | 84
Not Completed | 51 | 56
Not completed — Lack of Efficacy | 1 | 11
Not completed — Adverse Event | 31 | 20
Not completed — Physician Decision | 2 | 3
Not completed — Other - Unspecified | 8 | 14
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Ramipril: Participants were receiving CsA or TAC and either MMF, MPS, or AZA or steroids dosed per center's standard of care. Participants received ramipril 5 or 10 mg/d PO. 2-6 weeks after randomization, participants stopped TAC or CsA (within 21 days of SRL initiation) and received SRL, PO, 2-4 mg/d (6-12 mg on Day 1 if TAC or CsA withdrawn abruptly) to achieve target trough levels (7-15 ng/mL <1 year PT, 5-15 ng/mL ≥1 year PT) for up to 52 weeks. Ramipril was increased to 10-20 mg if U p/c was ≥0.5. If U p/c ≥0.5 persisted, losartan 50 mg/d was added; if U p/c ≥0.5 still persisted, losartan was increased to 100 mg/d. If then U p/c <0.5 was not maintained, study medication was discontinued and participant entered off-therapy phase of study.
- Total: Total of all reporting groups
Arm/Group | Ramipril | Placebo | Total
Number analyzed (Participants) | 155 | 140 | 295
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.8 (12.7) | 47.5 (12.9) | 47.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 50 | 98
  Male | 107 | 90 | 197

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had Initiated Losartan Therapy at 52 Weeks Following Conversion to SRL
Description: The event for each participant was defined as the initiation of losartan while on SRL and ramipril/placebo combination therapy. Participants who started losartan prior to SRL administration were not counted as events. Percentage was estimated using Kaplan-Meier method for time to event data.
Time Frame: From Day 1 of SRL conversion to 52 weeks after conversion
Population: Modified Intent to Treat (mITT) population: all participants in the safety population who took at least one dose of SRL.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 138 | 126
percentage of participants | 6.2 [2.7 to 11.6] | 23.2 [15.7 to 31.4]
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Test type: Superiority or Other; p = 0.0002, Log Rank — 2-sided p-value; alpha equals (=) 0.05; Stratified log-rank test with region and race strata; Hazard Ratio (HR) = 0.228, 95% CI 2-sided [0.099 to 0.528] — Stratified Cox proportional hazard model with region and race strata

2. Secondary Outcome: Percentage of Participants Who Had a Dose Escalation in Randomized Test Article (Ramipril or Placebo) by 52 Weeks Following Conversion to SRL
Description: Defined as the time from the first dose of SRL administration to the first dose escalation of randomized test article (ramipril or placebo; in weeks), or censored on the day that a participant stopped the combination of SRL and randomized test article (ramipril or placebo) if the participants did not experience any ramipril/placebo dose escalation following conversion to SRL. Dose-escalation was defined as an increase in total daily dose of ramipril/placebo compared to Day 1 post conversion. Percentage was estimated using Kaplan-Meier method for time to event data.
Time Frame: From Day 1 of SRL conversion to 52 weeks after conversion
Population: mITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 138 | 126
percentage of participants | 14.4 [8.7 to 21.3] | 29.2 [21.2 to 37.6]
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Test type: Superiority or Other; p = 0.0031, Log Rank — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); Stratified log-rank test with region and race strata; Hazard Ratio (HR) = 0.425, 95% CI 2-sided [0.237 to 0.763] — Stratified Cox proportional hazard model with region and race strata

3. Secondary Outcome: Percentage of Participants With U p/c <0.5 at 24 and 52 Weeks Following Conversion to Sirolimus
Description: Spot urine sample of protein and creatinine concentrations were obtained during the pre-SRL conversion period and after conversion.
Time Frame: 24 weeks and 52 weeks after conversion
Population: mITT population; includes assessments from On-Therapy and Off-Therapy Periods.
Measure: Number; unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 138 | 126
percentage of participants
  Up to 24 weeks post-conversion | 92.0 | 77.8
  Up to 52 weeks post-conversion | 82.6 | 73.0
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Up to 24 weeks post-conversion; Test type: Superiority or Other; p = 0.002, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 2: Comparison: Ramipril vs Placebo; Up to 52 weeks post-conversion; Test type: Superiority or Other; p = 0.074, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)

4. Secondary Outcome: Percentage of Participants With Urinary Albumin to Creatinine Ratio (U Alb/c) <0.5 at 24 and 52 Weeks Following Conversion to SRL
Description: Spot urine sample of albumin and creatinine concentrations were obtained during the pre-SRL conversion period and after conversion.
Time Frame: 24 weeks and 52 weeks after conversion
Population: mITT population; includes assessments from On-Therapy and Off-Therapy Periods.
Measure: Number; unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 138 | 126
percentage of participants
  Up to 24 weeks post-conversion | 95.7 | 89.7
  Up to 52 weeks post-conversion | 88.4 | 82.5
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Up to 24 weeks post-conversion; Test type: Superiority or Other; p = 0.093, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 2: Comparison: Ramipril vs Placebo; Up to 52 weeks post-conversion; Test type: Superiority or Other; p = 0.219, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)

5. Secondary Outcome: Percentage of Participants With Both U Alb/c <0.5 and U p/c <0.5 at 24 and 52 Weeks Following Conversion to SRL
Description: The U alb/c and U p/c must have been collected on the same day to be counted as the numerator.
Time Frame: 24 weeks and 52 weeks after conversion
Population: mITT population; includes assessments from On-Therapy and Off-Therapy Periods.
Measure: Number; unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 138 | 126
percentage of participants
  Up to 24 weeks post-conversion | 91.3 | 77.0
  Up to 52 weeks post-conversion | 79.0 | 70.6
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Up to 24 weeks post-conversion; Test type: Superiority or Other; p = 0.002, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 2: Comparison: Ramipril vs Placebo; Up to 52 weeks post-conversion; Test type: Superiority or Other; p = 0.121, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)

6. Secondary Outcome: U p/c at Baseline and Weeks 3, 4, 8, 12, 24, 30, 36, and 52 Following Conversion to SRL
Description: U p/c was measured in milligrams per milligram (mg/mg). The baseline U p/c values were the last values of the pre-SRL conversion period.
Time Frame: Baseline and 3, 4, 8, 12, 24, 30, 36, and 52 weeks after conversion
Population: mITT population; n (number) = number of participants assessed for the specified parameter at a given visit; only participants with nonmissing records of U p/c were included in the analysis. Includes measures collected from On-Therapy and Off-Therapy Periods.
Measure: Mean (Standard Deviation); unit: mg/mg
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 138 | 126
mg/mg
  Baseline (n=138,126) | 0.17 (0.37) | 0.15 (0.07)
  Week 3 (n=130,117) | 0.18 (0.11) | 0.23 (0.19)
  Week 4 (n=136,124) | 0.18 (0.09) | 0.28 (0.27)
  Week 8 (n=130,119) | 0.23 (0.39) | 0.31 (0.37)
  Week 12 (n=124,121) | 0.23 (0.30) | 0.38 (1.18)
  Week 24 (n=121,122) | 0.26 (0.40) | 0.31 (0.39)
  Week 30 (n=111,108) | 0.23 (0.23) | 0.32 (0.37)
  Week 36 (n=109,92) | 0.22 (0.13) | 0.29 (0.30)
  Week 52 (n=126,111) | 0.27 (0.31) | 0.35 (0.43)
Statistical Analysis 1: Comparison: Ramipril; Change from Baseline at Week 3, Ramipril; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.16 — Adjusted for baseline
Statistical Analysis 2: Comparison: Placebo; Change from Baseline at Week 3, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.36 — Adjusted for baseline
Statistical Analysis 3: Comparison: Ramipril vs Placebo; Change from baseline at Week 3, Ramipril versus (vs.) Placebo; Test type: Superiority or Other; p = 0.0098, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA model with change in the logarithmic Up/c as dependent variable, treatment and region/race as factors, and logarithmic baseline as covariate; Treatment Ratio = 0.85, 95% CI 2-sided [0.76 to 0.96] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change
Statistical Analysis 4: Comparison: Ramipril; Change from baseline at Week 4, Ramipril; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.18 — Adjusted for baseline
Statistical Analysis 5: Comparison: Placebo; Change from baseline at Week 4, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.52 — Adjusted for baseline
Statistical Analysis 6: Comparison: Ramipril vs Placebo; Change from baseline at Week 4, Ramipril vs. Placebo; Test type: Superiority or Other; p = 0.0003, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); [statistical method as in outcome 6, analysis 3]; Treatment Ratio = 0.78, 95% CI 2-sided [0.68 to 0.89] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change
Statistical Analysis 7: Comparison: Ramipril; Change from baseline at Week 8, Ramipirl; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.27 — Adjusted for baseline
Statistical Analysis 8: Comparison: Placebo; Change from baseline at Week 8, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.61 — Adjusted for baseline
Statistical Analysis 9: Comparison: Ramipril vs Placebo; Change from Baseline at Week 8, Ramipril vs. Placebo; Test type: Superiority or Other; p = 0.0016, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); [statistical method as in outcome 6, analysis 3]; Treatment Ratio = 0.79, 95% CI 2-sided [0.68 to 0.91] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change
Statistical Analysis 10: Comparison: Ramipril; Change from Baseline at Week 12, Ramipril; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.34 — Adjusted for baseline
Statistical Analysis 11: Comparison: Placebo; Change from Baseline at Week 12, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.63 — Adjusted for baseline
Statistical Analysis 12: Comparison: Ramipril vs Placebo; Change from Baseline at Week 12, Ramipril vs. Placebo; Test type: Superiority or Other; p = 0.0165, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); [statistical method as in outcome 6, analysis 3]; Treatment Ratio = 0.82, 95% CI 2-sided [0.70 to 0.96] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change
Statistical Analysis 13: Comparison: Ramipril; Change from Baseline at Week 24, Ramipril; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.48 — Adjusted for baseline
Statistical Analysis 14: Comparison: Placebo; Change from Baseline at Week 24, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.78 — Adjusted for baseline
Statistical Analysis 15: Comparison: Ramipril vs Placebo; Change from Baseline at Week 24, Ramipril vs. Placebo; Test type: Superiority or Other; p = 0.0264, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); [statistical method as in outcome 6, analysis 3]; Treatment Ratio = 0.83, 95% CI 2-sided [0.70 to 0.98] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change
Statistical Analysis 16: Comparison: Ramipril; Change from Baseline at Week 30, Ramipril; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.43 — Adjusted for baseline
Statistical Analysis 17: Comparison: Placebo; Change from Baseline at Week 30, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.82 — Adjusted for baseline
Statistical Analysis 18: Comparison: Ramipril vs Placebo; Change from Baseline at Week 30, Ramipril vs. Placebo; Test type: Superiority or Other; p = 0.0062, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); [statistical method as in outcome 6, analysis 3]; Treatment Ratio = 0.79, 95% CI 2-sided [0.66 to 0.93] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change
Statistical Analysis 19: Comparison: Ramipril; Change from Baseline at Week 36, Ramipril; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.40 — Adjusted for baseline
Statistical Analysis 20: Comparison: Placebo; Change from Baseline at Week 36, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.67 — Adjusted for baseline
Statistical Analysis 21: Comparison: Ramipril vs Placebo; Change from Baseline at Week 36, Ramipril vs. Placebo; Test type: Superiority or Other; p = 0.0341, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); [statistical method as in outcome 6, analysis 3]; Treatment Ratio = 0.84, 95% CI 2-sided [0.72 to 0.99] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change
Statistical Analysis 22: Comparison: Ramipril; Change from Baseline at Week 52, Ramipril; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.56 — Adjusted for baseline
Statistical Analysis 23: Comparison: Placebo; Change from Baseline at Week 52, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.86 — Adjusted for baseline
Statistical Analysis 24: Comparison: Ramipril vs Placebo; Change from Baseline at Week 52, Ramipril vs. Placebo; Test type: Superiority or Other; p = 0.0600, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); [statistical method as in outcome 6, analysis 3]; Treatment Ratio = 0.84, 95% CI 2-sided [0.70 to 1.01] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change

7. Secondary Outcome: U Alb/c at Baseline and Weeks 3, 4, 8, 12, 24, 30, 36, and 52 Following Conversion to SRL
Description: U alb/c was measured in mg/mg. Baseline U alb/c values were the last values of the pre-SRL conversion period.
Time Frame: Baseline and 3, 4, 8, 12, 24, 30, 36, and 52 weeks after conversion
Population: mITT population; n=number of participants assessed for the specified parameter at a given visit; only participants with nonmissing records of U alb/c were included in the analysis. Includes measures collected from On-Therapy and Off-Therapy Periods.
Measure: Mean (Standard Deviation); unit: mg/mg
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 138 | 126
mg/mg
  Baseline (n=138,126) | 0.04 (0.26) | 0.02 (0.02)
  Week 3 (n=129,117) | 0.03 (0.05) | 0.06 (0.11)
  Week 4 (n=136,124) | 0.03 (0.04) | 0.09 (0.16)
  Week 8 (n=129,119) | 0.06 (0.31) | 0.11 (0.24)
  Week 12 (n=124,121) | 0.05 (0.09) | 0.17 (0.84)
  Week 24 (n=121,122) | 0.08 (0.24) | 0.11 (0.28)
  Week 30 (n=111,108) | 0.06 (0.13) | 0.11 (0.21)
  Week 36 (n=109,92) | 0.05 (0.08) | 0.10 (0.21)
  Week 52 (n=126,111) | 0.09 (0.21) | 0.15 (0.31)
Statistical Analysis 1: Comparison: Ramipril; Change from Baseline at Week 3, Ramipril; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.46 — Adjusted for baseline
Statistical Analysis 2: Comparison: Placebo; Change from Baseline at Week 3, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 2.05 — Adjusted for baseline
Statistical Analysis 3: Comparison: Ramipril vs Placebo; Change from Baseline at Week 3, Ramipril vs. Placebo; Test type: Superiority or Other; p = 0.0034, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA model with change in the logarithmic U alb/c as dependent variable, treatment and region/race as factors, and logarithmic baseline as covariate; Treatment Ratio = 0.71, 95% CI 2-sided [0.57 to 0.89] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change
Statistical Analysis 4: Comparison: Ramipril; Change from Baseline at Week 4, Ramipril; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.43 — Adjusted for baseline
Statistical Analysis 5: Comparison: Placebo; Change from Baseline at Week 4, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 2.37 — Adjusted for baseline
Statistical Analysis 6: Comparison: Ramipril vs Placebo; Change from Baseline at Week 4, Ramipril vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); [statistical method as in outcome 7, analysis 3]; Treatment Ratio = 0.60, 95% CI 2-sided [0.47 to 0.76] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change
Statistical Analysis 7: Comparison: Ramipril; Change from Baseline at Week 8, Ramipril; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.67 — Adjusted for baseline
Statistical Analysis 8: Comparison: Placebo; Change from Baseline at Week 8, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 2.74 — Adjusted for baseline
Statistical Analysis 9: Comparison: Ramipril vs Placebo; Change from Baseline at Week 8, Ramipril vs. Placebo; Test type: Superiority or Other; p = 0.0002, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); [statistical method as in outcome 7, analysis 3]; Treatment Ratio = 0.61, 95% CI 2-sided [0.47 to 0.79] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change
Statistical Analysis 10: Comparison: Ramipril; Change from Baseline at Week 12, Ramipril; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 1.91 — Adjusted for baseline
Statistical Analysis 11: Comparison: Placebo; Change from Baseline at Week 12, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 2.92 — Adjusted for baseline
Statistical Analysis 12: Comparison: Ramipril vs Placebo; Change from Baseline at Week 12, Ramipril vs. Placebo; Test type: Superiority or Other; p = 0.0032, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); [statistical method as in outcome 7, analysis 3]; Treatment Ratio = 0.65, 95% CI 2-sided [0.49 to 0.87] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change
Statistical Analysis 13: Comparison: Ramipril; Change from Baseline at Week 24, Ramipril; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 2.33 — Adjusted for baseline
Statistical Analysis 14: Comparison: Placebo; Change from Baseline at Week 24, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 3.39 — Adjusted for baseline
Statistical Analysis 15: Comparison: Ramipril vs Placebo; Change from Baseline at Week 24, Ramipril vs. Placebo; Test type: Superiority or Other; p = 0.0130, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); [statistical method as in outcome 7, analysis 3]; Treatment Ratio = 0.69, 95% CI 2-sided [0.51 to 0.92] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change
Statistical Analysis 16: Comparison: Ramipril; Change from Baseline at Week 30, Ramipril; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 2.50 — Adjusted for baseline
Statistical Analysis 17: Comparison: Placebo; Change from Baseline at Week 30, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 3.39 — Adjusted for baseline
Statistical Analysis 18: Comparison: Ramipril vs Placebo; Change from Baseline at Week 30, Ramipril vs. Placebo; Test type: Superiority or Other; p = 0.0577, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); [statistical method as in outcome 7, analysis 3]; Treatment Ratio = 0.74, 95% CI 2-sided [0.54 to 1.01] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change
Statistical Analysis 19: Comparison: Ramipril; Change from Baseline at Week 36, Ramipril; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 2.52 — Adjusted for baseline
Statistical Analysis 20: Comparison: Placebo; Change from Baseline at Week 36, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 3.27 — Adjusted for baseline
Statistical Analysis 21: Comparison: Ramipril vs Placebo; Change from Baseline at Week 36, Ramipril vs. Placebo; Test type: Superiority or Other; p = 0.1146, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); [statistical method as in outcome 7, analysis 3]; Treatment Ratio = 0.77, 95% CI 2-sided [0.56 to 1.07] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change
Statistical Analysis 22: Comparison: Ramipril; Change from Baseline at Week 52, Ramipril; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 2.92 — Adjusted for baseline
Statistical Analysis 23: Comparison: Placebo; Change from Baseline at Week 52, Placebo; Test type: Superiority or Other; Adjusted Geometric Mean Fold Change = 3.45 — Adjusted for baseline
Statistical Analysis 24: Comparison: Ramipril vs Placebo; Change from Baseline at Week 52, Ramipril vs. Placebo; Test type: Superiority or Other; p = 0.3496, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); [statistical method as in outcome 7, analysis 3]; Treatment Ratio = 0.85, 95% CI 2-sided [0.60 to 1.20] — Treatment ratio (Ramipril/Placebo) in the geometric mean fold-change

8. Secondary Outcome: Percentage of Participants Who Discontinued SRL Therapy at 24 and 52 Weeks Following Conversion to SRL
Description: Defined as the percentage of participants who stop SRL (as test article) between the first day of SRL and either Week 24 or Week 52 following conversion to SRL. If a participant had a >14 day gap in SRL use, the stop date of SRL was the date of the last SRL use before it was re-initiated. Participants who early terminate SRL at Week 24 were defined as having SRL stop day less than or equal to (≤) Day 190 (selected as the midpoint between Weeks 24 and 30). Participants who early terminate SRL at Week 52 were defined as having SRL stop day ≤Day 337 (selected as the midpoint between Weeks 44 and 52).
Time Frame: 24 weeks and 52 weeks after conversion
Population: mITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 138 | 126
percentage of participants
  Up to 24 weeks post-conversion | 15.2 | 15.9
  Up to 52 weeks post-conversion | 19.6 | 28.6
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Up to 24 weeks post-conversion; Test type: Superiority or Other; p = 1.0000, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 2: Comparison: Ramipril vs Placebo; Up to 52 weeks post-conversion; Test type: Superiority or Other; p = 0.1115, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)

9. Secondary Outcome: Abbreviated Modified Diet in Renal Disease (MDRD) Glomerular Filtration Rate (GFR) at Weeks 12, 24, and 52 Following Conversion to SRL
Description: Calculated in millimeters per minute per 1.73 square meters (mL/min/1.73m^2). Age and corresponding creatinine at each visit (Weeks 12, 24, and 52) were used to calculate GFR.
Time Frame: 12, 24, and 52 weeks following conversion
Population: mITT population; n=number of participants assessed for the specified parameter at a given visit. Includes measures collected from On-Therapy and Off-Therapy Periods.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 138 | 126
mL/min/1.73 m^2
  Baseline (n=138,126) | 62.06 (14.08) | 63.30 (15.64)
  Week 12 (n=125,122) | 64.91 (16.54) | 66.58 (15.26)
  Week 24 (n=123,122) | 65.18 (17.99) | 63.85 (16.49)
  Week 52 (n=128,115) | 64.17 (16.79) | 63.41 (15.54)
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Change from Baseline at Week 12; Test type: Superiority or Other; p = 0.4933, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA model with MDRD change as dependent variable, treatment and region/race as factors, and baseline as covariate; Adjusted LS Mean Difference = -0.86, 95% CI 2-sided [-3.33 to 1.61], Standard Error of Mean 1.26 — Adjusted for baseline
Statistical Analysis 2: Comparison: Ramipril vs Placebo; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.0888, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA model with MDRD change as dependent variable, treatment and region/race as factors, and baseline as covariate; Adjusted LS Mean Difference = 2.48, 95% CI 2-sided [-0.38 to 5.33], Standard Error of Mean 1.45 — Adjusted for baseline
Statistical Analysis 3: Comparison: Ramipril vs Placebo; Change from Baseline at Week 52; Test type: Superiority or Other; p = 0.1475, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA model with MDRD change as dependent variable, treatment and region/race as factors, and baseline as covariate; Adjusted LS Mean Difference = 2.12, 95% CI 2-sided [-0.75 to 4.99], Standard Error of Mean 1.46 — Adjusted for baseline

10. Secondary Outcome: Fraction of Albumin (Milligrams Per Deciliter [mg/dL]) to Protein (mg/dL) in Urine at 24 and 52 Weeks After Conversion to SRL
Description: Baseline fraction was the last value of the pre-SRL conversion period. Only the last value of U p/c or U alb/c was used for analysis if multiple measurements occurred in the same data anlysis interval. Fraction of albumin and protein was calculated only when urine protein was 6.2 mg/dL or higher. For urine albumin, if the value was reported as '<xx.x', the numerical portion of the value was used in the calculation of fraction of albumin and protein.
Time Frame: 24 weeks and 52 weeks after conversion
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: (mg/dL)/(mg/dL)
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 111 | 110
(mg/dL)/(mg/dL)
  Week 24 (n=104,110) | 0.19 (0.17) | 0.25 (0.19)
  Week 52 (n=111,105) | 0.22 (0.18) | 0.25 (0.20)
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Week 24; Test type: Superiority or Other; p = 0.1167, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); Log (Fraction of albumin to protein in urine) as dependent variable, treatment and region/race as factor, and Log(baseline) as covariate; Treatment Ratio = 0.84, 95% CI 2-sided [0.68 to 1.04] — Treatment ratio (Ramipril/Placebo) in the geometric mean
Statistical Analysis 2: Comparison: Ramipril vs Placebo; Week 52; Test type: Superiority or Other; p = 0.7519, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); [statistical method as in outcome 10, analysis 1]; Treatment Ratio = 1.04, 95% CI 2-sided [0.82 to 1.31] — Treatment ratio (Ramipril/Placebo) in the geometric mean

11. Secondary Outcome: Percentage of Participants With Potentially Clinically Important Blood Pressure (BP) Values by Diastolic and Systolic BP Category
Description: BP values of potential clinical importance were recorded and categorized as follows: diastolic BP (DBP) ≤50 millimeters of mercury (mmHg) or ≥110 mmHg and systolic BP (SBP) ≤90 mmHg and ≥180 mmHg. Data were summarized for the on-therapy period and the off-therapy period and for the pre-SRL period.
Time Frame: Baseline, Pre-SRL (from first dose of ramipril/placebo up to SRL conversion), On-Therapy (up to 52 weeks after SRL conversion), and Off-Therapy Period (up to 56 weeks after SRL conversion)
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 155 | 140
percentage of participants
  Baseline, Low DBP ≤50 mmHg (n=155,140) | 0.0 | 0.7
  Baseline, Low SBP: ≤90 mmHg (n=155,140) | 0.0 | 0.7
  Pre-SRL, Low DBP: ≤50 mmHg (n=152,135) | 0.0 | 0.7
  Pre-SRL, High DBP: ≥110 mmHg (n=152,135) | 0.0 | 1.5
  Pre-SRL, Low SBP: ≤90 mmHg (n=152,135) | 0.0 | 0.7
  Pre-SRL, High SBP: ≥180 mmHg (n=152,135) | 0.7 | 0.7
  On Therapy, Low DBP: ≤50 mmHg (n=138,126) | 3.6 | 2.4
  On Therapy, High DBP: ≥110 mmHg (n=138,126) | 0.0 | 1.6
  On Therapy, Low SBP: ≤90 mmHg (n=138,126) | 3.6 | 4.0
  On Therapy, High SBP: ≥180 mmHg (n=138,126) | 0.7 | 4.0
  Off Therapy, High DBP ≥110 mmHg (n=35,69) | 2.9 | 1.4
  Off Therapy, Low SBP: ≤90 mmHg (n=35,69) | 2.9 | 1.4
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Pre-SRL, Low DBP ≤50 mmHg; Test type: Superiority or Other; p = 0.470, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 2: Comparison: Ramipril vs Placebo; Pre-SRL, High DBP ≥110 mmHg; Test type: Superiority or Other; p = 0.220, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 3: Comparison: Ramipril vs Placebo; Pre-SRL, Low SBP: ≤90 mmHg; Test type: Superiority or Other; p = 0.470, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 4: Comparison: Ramipril vs Placebo; Pre-SRL, High SBP: ≥180 mmHg; Test type: Superiority or Other; p = 1.000, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 5: Comparison: Ramipril vs Placebo; On Therapy, Low DBP ≤50 mmHg; Test type: Superiority or Other; p = 0.725, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 6: Comparison: Ramipril vs Placebo; On Therapy, High DBP ≥110 mmHg; Test type: Superiority or Other; p = 0.227, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 7: Comparison: Ramipril vs Placebo; On Therapy, Low SBP: ≤90 mmHg; Test type: Superiority or Other; p = 1.000, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 8: Comparison: Ramipril vs Placebo; On Therapy, High SBP: ≥180 mmHg; Test type: Superiority or Other; p = 0.106, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 9: Comparison: Ramipril vs Placebo; Off Therapy, High DBP ≥110 mmHg; Test type: Superiority or Other; p = 1.000, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 10: Comparison: Ramipril vs Placebo; Off Therapy, Low SBP: ≤90 mmHg; Test type: Superiority or Other; p = 1.000, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 11: Comparison: Ramipril vs Placebo; Baseline, Low DBP ≤50 mmHg; Test type: Superiority or Other; p = 0.475, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 12: Comparison: Ramipril vs Placebo; Baseline, Low SBP: ≤90 mmHg; Test type: Superiority or Other; p = 0.475, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)

12. Secondary Outcome: SRL Time-Normalized Trough Concentration (Cmin,TN) by Time Interval
Description: Cmin,TN was determined for SRL using the area method for the intervals: 0-2 weeks, >2-4 weeks, >4-12 weeks, >12-24 weeks, >24-36 weeks and >36-52 weeks using the equation:Cmin,TN = AUCi-j/timej-timeiwhere AUC is the area under the concentration-time curve, i is the beginning of the interval and j is the end of the interval. Cmin,TN was calculated for participants who did not dropout of studies, but were missing concentrations at the interval endpoints by carrying the last observed concentration forward to the interval endpoint.
Time Frame: From Day 1 of SRL conversion to 52 weeks after conversion
Population: Safety population; n=number of participants assessed for the specified parameter for the given time interval; only participants dosed throughout the interval were included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ramipril
Number analyzed (Participants) | 258
ng/mL
  0-2 weeks (n=258) | 9.853 (6.0250)
  >2-4 weeks (n=257) | 9.872 (4.1408)
  >4-12 weeks (n=256) | 9.273 (3.1763)
  >12-24 weeks (n=244) | 9.274 (2.8944)
  >24-36 weeks (n=226) | 9.316 (3.1535)
  >36-52 weeks (n=193) | 8.961 (2.9031)
  0-52 weeks (n=264) | 9.300 (2.2678)

13. Secondary Outcome: Percentage of Participants With Hemoglobin Levels ≤100 Grams Per Liter (g/L)
Time Frame: as for outcome 11
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 155 | 140
percentage of participants
  Baseline (n=155,140) | 1.3 | 1.4
  Pre-SRL (n=148,129) | 2.0 | 0.8
  On-Therapy (n=138,124) | 17.4 | 12.1
  Off-Therapy (n=33,34) | 9.1 | 2.9
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Baseline; Test type: Superiority or Other; p = 1.000, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 2: Comparison: Ramipril vs Placebo; Pre-SRL; Test type: Superiority or Other; p = 0.626, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 3: Comparison: Ramipril vs Placebo; On-Therapy; Test type: Superiority or Other; p = 0.297, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 4: Comparison: Ramipril vs Placebo; Off-Therapy; Test type: Superiority or Other; p = 0.356, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)

14. Secondary Outcome: Percentage of Participants Using Red Blood Cell Production Stimulants (Erythropoiesis Stimulating Agents [ESAs])
Time Frame: as for outcome 11
Population: Safety population; n=number of participants analyzed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 155 | 140
percentage of participants
  Baseline (n=155,140) | 5.8 | 1.4
  Pre-SRL (n=155,140) | 4.5 | 0.7
  On-Therapy (n=138,126) | 4.3 | 3.2
  Off-Therapy (n=136,122) | 1.5 | 4.1
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Baseline; Test type: Superiority or Other; p = 0.064, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 2: Comparison: Ramipril vs Placebo; Pre-SRL; Test type: Superiority or Other; p = 0.069, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 3: Comparison: Ramipril vs Placebo; On-Therapy; Test type: Superiority or Other; p = 0.752, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 4: Comparison: Ramipril vs Placebo; Off-Therapy; Test type: Superiority or Other; p = 0.261, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)

15. Secondary Outcome: Change From Baseline in Fasting Lipid Parameters (Millimoles Per Liter [mmol/L]) at 4, 12, 24, and 52 Weeks Following Conversion to SRL
Description: Parameters assessed included (all fasting) total cholesterol (TC), triglycerides, low-density lipoprotein cholesterol (LDL-C), high-densitylipoprotein cholesterol (HDL-C).
Time Frame: 4, 12, 24, and 52 weeks after conversion
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 128 | 109
mmol/L
  TC, Week 4 (n=128,109) | 0.83 (0.06) | 0.91 (0.09)
  TC, Week 12 (n=115,108) | 0.94 (0.09) | 0.92 (0.10)
  TC, Week 24 (n=105,102) | 0.91 (0.12) | 0.87 (0.09)
  TC, Week 52 (n=94,79) | 0.84 (0.11) | 0.69 (0.12)
  HDL-C, Week 4 (n=125,107) | 0.06 (0.02) | 0.09 (0.03)
  HDL-C, Week 12 (n=114,104) | 0.03 (0.02) | 0.03 (0.02)
  HDL-C, Week 24 (n=102,100) | 0.07 (0.03) | 0.04 (0.03)
  HDL-C, Week 52 (n=92,78) | 0.12 (0.03) | 0.06 (0.04)
  LDL-C, Week 4 (n=123,100) | 0.59 (0.06) | 0.56 (0.07)
  LDL-C, Week 12 (n=109,96) | 0.66 (0.08) | 0.53 (0.08)
  LDL-C, Week 24 (n=96,95) | 0.66 (0.10) | 0.56 (0.08)
  LDL-C, Week 52 (n=90,73) | 0.56 (0.10) | 0.27 (0.09)
  Triglycerides, Week 4 (n=127,108) | 0.41 (0.07) | 0.65 (0.10)
  Triglycerides, Week 12 (n=114,107) | 0.59 (0.10) | 0.79 (0.11)
  Triglycerides, Week 24 (n=104,102) | 0.54 (0.11) | 0.72 (0.13)
  Triglycerides, Week 52 (n=93,77) | 0.44 (0.10) | 0.58 (0.14)
Statistical Analysis 1: Comparison: Ramipril vs Placebo; TC, Week 4; Test type: Superiority or Other; p = 0.381, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = -0.09, Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Ramipril vs Placebo; TC, Week 12; Test type: Superiority or Other; p = 0.956, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = 0.01, Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Ramipril vs Placebo; TC, Week 24; Test type: Superiority or Other; p = 0.903, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in adjusted means = 0.02, Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: Ramipril vs Placebo; TC, Week 52; Test type: Superiority or Other; p = 0.503, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = 0.10, Standard Error of Mean 0.15
Statistical Analysis 5: Comparison: Ramipril vs Placebo; HDL-C, Week 4; Test type: Superiority or Other; p = 0.451, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = -0.03, Standard Error of Mean 0.03
Statistical Analysis 6: Comparison: Ramipril vs Placebo; HDL-C, Week 12; Test type: Superiority or Other; p = 0.919, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = -0.00, Standard Error of Mean 0.03
Statistical Analysis 7: Comparison: Ramipril vs Placebo; HDL-C, Week 24; Test type: Superiority or Other; p = 0.637, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = 0.02, Standard Error of Mean 0.04
Statistical Analysis 8: Comparison: Ramipril vs Placebo; HDL-C, Week 52; Test type: Superiority or Other; p = 0.229, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = 0.05, Standard Error of Mean 0.05
Statistical Analysis 9: Comparison: Ramipril vs Placebo; LDL-C, Week 4; Test type: Superiority or Other; p = 0.766, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = 0.03, Standard Error of Mean 0.09
Statistical Analysis 10: Comparison: Ramipril vs Placebo; LDL-C, Week 12; Test type: Superiority or Other; p = 0.217, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = 0.14, Standard Error of Mean 0.11
Statistical Analysis 11: Comparison: Ramipril vs Placebo; LDL-C, Week 24; Test type: Superiority or Other; p = 0.457, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = 0.10, Standard Error of Mean 0.13
Statistical Analysis 12: Comparison: Ramipril vs Placebo; LDL-C, Week 52; Test type: Superiority or Other; p = 0.041, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = 0.26, Standard Error of Mean 0.13
Statistical Analysis 13: Comparison: Ramipril vs Placebo; Triglycerides, Week 4; Test type: Superiority or Other; p = 0.044, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = -0.25, Standard Error of Mean 0.12
Statistical Analysis 14: Comparison: Ramipril vs Placebo; Triglycerides, Week 12; Test type: Superiority or Other; p = 0.180, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = -0.20, Standard Error of Mean 0.15
Statistical Analysis 15: Comparison: Ramipril vs Placebo; Triglycerides, Week 24; Test type: Superiority or Other; p = 0.264, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = -0.19, Standard Error of Mean 0.17
Statistical Analysis 16: Comparison: Ramipril vs Placebo; Triglycerides, Week 52; Test type: Superiority or Other; p = 0.408, ANCOVA — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); ANCOVA with treatment as a factor and baseline as a covariate; Difference in Adjusted Means = -0.14, Standard Error of Mean 0.17

16. Secondary Outcome: Biopsy-Confirmed Acute Rejection (BCAR) - Number of Participants With an Event
Description: BCAR was defined according to updated Banff criteria (1997)for renal allograft rejection. The time to the first BCAR was defined as the date of first BCAR to the date of the first dose of SRL (in weeks). Participants without BCAR were censored at the time of withdrawal from the study.
Time Frame: From Day 1 of SRL conversion to 52 weeks after conversion
Population: mITT population; includes BCAR occurring in On-Therapy and Off-Therapy Periods.
Measure: Number; unit: participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 138 | 126
participants | 13 | 5
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Test type: Superiority or Other; p = 0.0732, Log Rank — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); Hazard Ratio (HR) = 2.487, 95% CI 2-sided [0.887 to 6.978] — Hazard ratio was based on the Cox proportional hazards model

17. Secondary Outcome: Percentage of Participants With First BCAR at 24 and 52 Weeks Following Conversion to SRL
Description: BCAR was defined according to updated Banff criteria (1997)for renal allograft rejection. Participants without BCAR were censored at the time of withdrawal from the study. Defined as the first BCAR occurring on therapy following conversion to SRL based on the mITT population. Time to first BCAR was defined as the date of first BCAR to date of the first dose of SRL (in weeks). Percentages were estimated using the Kaplan-Meier method for time to event data.
Time Frame: 24 weeks and 52 weeks after conversion
Population: mITT population; includes BCAR occurring in the On-Therapy and Off-Therapy Periods
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 138 | 126
percentage of participants
  24 weeks post-conversion | 8.0 [4.2 to 13.3] | 0.8 [0.1 to 4.0]
  52 weeks post-conversion | 9.5 [5.3 to 15.1] | 3.2 [1.1 to 7.5]

18. Secondary Outcome: Number of Participants With BCAR by Severity of First BCAR
Description: Severity was summarized by type (antibody versus T-cell) and by phase: post-SRL (where both on-therapy and off-therapy events are included) and post-SRL (on-therapy). BCAR was categorized using Banff criteria as antibody-mediated (AM) or T-cell. AM BCAR severity was graded as Grade I (mild), Grade II (moderate [mod]), and Grade III (severe). T-cell BCAR severity was graded as 'Grade Ia, Ib (mild), Grade IIa, IIb (mod), and Grade III (severe). If a participant had both T-cell BCAR and antibody-mediated BCAR on the first rejection, the participant was counted in each category. For participants with T-cell BCAR (post-SRL and post-SRL On -Therapy) the p-value could not be calculated and all events were mild in severity.
Time Frame: From Day 1 of SRL conversion to 52 weeks after conversion
Population: mITT population; only participants with BCAR were included in the anlaysis.
Measure: Number; unit: participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 13 | 8
participants
  Post-SRL, AM BCAR, Grade I (mild) | 1 | 2
  Post-SRL, AM BCAR, Grade II (mod) | 0 | 1
  Post-SRL, AM BCAR, Grade III (severe) | 0 | 1
  Post-SRL, T-Cell BCAR, Grade I (mild) | 12 | 4
  Post-SRL (On-Therapy), AM BCAR, Grade I (mild) | 1 | 1
  Post-SRL (On-Therapy), AM BCAR, Grade II (mod) | 0 | 1
  Post-SRL (On-Therapy), T-Cell BCAR, Grade I (mild) | 10 | 3
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Post-SRL, AM BCAR; Test type: Superiority or Other; p = 0.7165, Cochran-Mantel-Haenszel — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); Cochran-Mantel-Haenszel row mean test
Statistical Analysis 2: Comparison: Ramipril vs Placebo; Post-SRL (On-Therapy), AM BCAR; Test type: Superiority or Other; p = 0.4795, Cochran-Mantel-Haenszel — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity); Cochran-Mantel-Haenszel row mean test

19. Secondary Outcome: Percentage of Participants With Graft Loss at 24 and 52 Weeks Following Conversion to SRL
Description: Graft loss was defined as physical loss (nephrectomy orretransplantation), functional loss (requiring dialysis for ≥56days with no return of graft function), or death.
Time Frame: 24 weeks and 52 weeks after conversion
Population: mITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 138 | 126
percentage of participants
  Week 24 | 0.0 | 0.0
  Week 52 | 0.0 | 0.8
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Week 52; Test type: Superiority or Other; p = 0.4773, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)

20. Secondary Outcome: Percentage of Participants Using Statins
Time Frame: as for outcome 11
Population: Safety population; n=number of participants analyzed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 155 | 140
percentage of participants
  Baseline (n=155,140) | 45.8 | 36.4
  Pre-SRL (n=155,140) | 45.2 | 40.0
  On-Therapy (n=138,126) | 67.4 | 72.2
  Off-Therapy (n=136,122) | 62.5 | 68.9
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Baseline; Test type: Superiority or Other; p = 0.124, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 2: Comparison: Ramipril vs Placebo; Pre-SRL; Test type: Superiority or Other; p = 0.410, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 3: Comparison: Ramipril vs Placebo; On-Therapy; Test type: Superiority or Other; p = 0.423, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 4: Comparison: Ramipril vs Placebo; Off-Therapy; Test type: Superiority or Other; p = 0.297, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)

21. Secondary Outcome: Percentage of Participants With an Infection
Description: Includes treatment-emergent adverse events based on categorization by the investigator as 'infection', regardless of the event preferred term in Medical Dictionary for Regulatory Activities (MedDRA.)
Time Frame: From Day 1 of Ramipril/Placebo to 52 weeks after SRL conversion
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 155 | 140
percentage of participants | 54.2 | 56.4
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Test type: Superiority or Other; p = 0.726, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)

22. Secondary Outcome: Percentage of Participants With Angioedema
Description: Includes treatment-emergent adverse events based on categorization by the investigator as angioedema, regardless of the event preferred term in MedDRA.
Time Frame: From Day 1 of Ramipril/Placebo to 52 weeks after SRL conversion
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 155 | 140
percentage of participants | 1.3 | 1.4
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Test type: Superiority or Other; p = 1.000, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)

23. Secondary Outcome: Percentage of Participants With Malignancy
Description: Includes treatment-emergent adverse events based on categorization by the investigator as 'malignancy', regardless of the event preferredterm in MedDRA.
Time Frame: From Day 1 of Ramipril/Placebo to 52 weeks after SRL conversion
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 155 | 140
percentage of participants | 3.9 | 2.9
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Test type: Superiority or Other; p = 0.753, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)

24. Secondary Outcome: Percentage of Participants With Hyperkalemia
Description: Hyperkalemia defined as serum potassium >5.6 millimoles per liter (mmol/L)
Time Frame: as for outcome 11
Population: Safety population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 155 | 140
percentage of participants
  Baseline (n=155,140) | 0.0 | 1.4
  Pre-SRL (n=151,135) | 4.6 | 1.5
  On-Therapy (n=138,124) | 0.7 | 1.6
  Off-Therapy (n=34,36) | 2.9 | 0.0
Statistical Analysis 1: Comparison: Ramipril vs Placebo; Baseline; Test type: Superiority or Other; p = 0.224, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 2: Comparison: Ramipril vs Placebo; Pre-SRL; Test type: Superiority or Other; p = 0.179, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 3: Comparison: Ramipril vs Placebo; On-Therapy; Test type: Superiority or Other; p = 0.604, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)
Statistical Analysis 4: Comparison: Ramipril vs Placebo; Off-Therapy; Test type: Superiority or Other; p = 0.486, Fisher Exact — 2-sided p-value; alpha=0.05 (unadjusted for multiplicity)

ADVERSE EVENTS:
Time Frame: Randomization through Week 52 following conversion to SRL
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Ramipril | Placebo
Serious Adverse Events (participants affected / at risk) | 50/155 | 39/140
Other Adverse Events (participants affected / at risk) | 134/155 | 123/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ramipril (N=155) | Placebo (N=140)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Haemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 2
Embolism (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Superior vena caval stenosis (Vascular disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Chest pain (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Kidney transplant rejection (Immune system disorders) | 3 | 3
Transplant rejection (Immune system disorders) | 11 | 1
Cellulitis (Infections and infestations) | 4 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1
H1N1 influenza (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Herpes zoster disseminated (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Oral bacterial infection (Infections and infestations) | 1 | 0
Oral infection (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 1
Viral infection (Infections and infestations) | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 1
Graft complication (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Medication error (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 2 | 1
Blood urea increased (Investigations) | 1 | 0
Clostridium test positive (Investigations) | 0 | 1
Cytomegalovirus test positive (Investigations) | 1 | 0
Immunosuppressant drug level increased (Investigations) | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Renal cyst ruptured (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Syncope (Nervous system disorders) | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ramipril (N=155) | Placebo (N=140)
Anaemia (Blood and lymphatic system disorders) | 18 | 10
Leukopenia (Blood and lymphatic system disorders) | 19 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 12
Hypertension (Vascular disorders) | 10 | 14
Hypotension (Vascular disorders) | 14 | 7
Aphthous stomatitis (Gastrointestinal disorders) | 12 | 14
Diarrhoea (Gastrointestinal disorders) | 40 | 37
Mouth ulceration (Gastrointestinal disorders) | 12 | 17
Nausea (Gastrointestinal disorders) | 8 | 9
Stomatitis (Gastrointestinal disorders) | 7 | 11
Vomiting (Gastrointestinal disorders) | 10 | 8
Fatigue (General disorders) | 12 | 7
Local swelling (General disorders) | 3 | 9
Oedema peripheral (General disorders) | 27 | 30
Pyrexia (General disorders) | 11 | 9
Bronchitis (Infections and infestations) | 4 | 7
Nasopharyngitis (Infections and infestations) | 8 | 7
Upper respiratory tract infection (Infections and infestations) | 27 | 16
Urinary tract infection (Infections and infestations) | 12 | 13
Blood creatinine increased (Investigations) | 24 | 11
Weight increased (Investigations) | 8 | 5
Proteinuria (Renal and urinary disorders) | 8 | 15
Dyslipidaemia (Metabolism and nutrition disorders) | 14 | 19
Hypercholesterolaemia (Metabolism and nutrition disorders) | 17 | 14
Hyperlipidaemia (Metabolism and nutrition disorders) | 15 | 9
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 16 | 15
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 9
Dizziness (Nervous system disorders) | 12 | 10
Headache (Nervous system disorders) | 19 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 12
Acne (Skin and subcutaneous tissue disorders) | 18 | 25
Rash (Skin and subcutaneous tissue disorders) | 5 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.